CLINICAL TRIAL: NCT01521130
Title: Imaging the Effect of Centrotemporal Spikes and Seizures on Language in Children
Acronym: FIRST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS065840-01 (NIH); R01NS065840-01 (NIH)
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Benign Childhood Epilepsy With Centro-Temporal Spikes
Keywords: Benign Childhood Epilepsy With Centrotemporal Spikes; Benign Rolandic Epilepsy
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Control (No Intervention): Healthy Control
- BECTS, no medication (No Intervention): BECTS, no medication
- Levetiracetam Higher dose (Experimental): Levetiracetam Higher dose
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Medication doses are defined on a mg/kg basis. Dosage form, frequency and titration schedule is based on accepted clinical practice.
  Other Names: Keppra
  Arms: Levetiracetam Higher dose

SUMMARY:
This project examines how seizures, and abnormal brain activity, affect language skill in children with Benign Childhood Epilepsy with Centro-Temporal Spikes (BECTS). BECTS is a common type of childhood epilepsy, and while BECTS patients stop having seizures by their late teenage years, many studies have shown that these children have language problems that may lead to academic and social difficulties. Using standardized language testing, monitoring of brain activity, and MRI brain imaging, this project aims to determine what particular combination of BECTS symptoms put children most at risk for language problems and whether treatment with anti-epileptic medications may be helpful.

DETAILED DESCRIPTION:
Benign Childhood Epilepsy with Centro-Temporal Spikes (BECTS), an extremely common type of childhood epilepsy, is traditionally assumed to have a benign course, but recent studies have shown that cognitive function, especially language, is often impaired in BECTS patients. However, it is not clear whether ithe seizures, the centrotemporal spikes (CTS), or other factors cause the negative cognitive consequences that may impact school performance and social interaction. BECTS patients have scattered seizures but very frequent CTS, and may be suffering with undiagnosed cognitive and language deficits. This suggests a causal role for CTS that has not yet been investigated in detail. This project will examine the impact of seizures and CTS on neurocognitive function in BECTS patients, at diagnosis and after one year. We will gather critical information regarding the effect of the anti-epileptic medication levetiracetam on CTS, which will inform a future Phase III clinical trial aimed at eliminating CTS and improving long term outcome.

This study will explore the interactions between CTS, seizures and neuropsychological outcomes using Functional MRI of language in order to decipher changes in neural circuitry that underlie language deficits found in children with BECTS. Using standardized neuropsychological testing and fMRI at the time of diagnosis, this study will first characterize the nature and incidence of language problems in children with BECTS, separating the effects of CTS and seizures. It is expected that children with BECTS will perform below normative standards on tests of language skill, accompanied by aberrations in the neural circuitry supporting language processing as tested with fMRI. These data will also make it possible to characterize which children with BECTS are most at risk for language problems, by taking into account contributing factors such as number of seizures, age of onset, and frequency and lateralization of CTS.

The proposed exploratory clinical trial will also provide key information needed to properly design and conduct a future double blind Phase III randomized clinical trial (RCT) children aimed at improving language outcome through elimination of CTS. Using an open-label dose-ranging design and 1-year follow up, we will determine the best dose of levetiracetam to control seizures, eliminate CTS and be well tolerated. We will also examine the extent of changes in language function and neural circuitry of language with 1-year follow-up neuropsychological testing and fMRI in LEV-treated and untreated BECTS compared to controls (which will document the natural history of neuropsychological function in untreated BECTS children and give additional information about the effect of LEV). The current study will provide crucial information for a future double blind RCT that will the compare the selected dose of levetiracetam to carbamazepine (the current standard of care) in BECTS. This would change clinical practice by demonstrating the need for AED treatment in BECTS to eliminate CTS, in turn improving long term language and cognitive outcome.

ELIGIBILITY:
Inclusion Criteria for BECTS participants

Diagnosis: Child has newly diagnosed BECTS according to International League Against Epilepsy (ILAE) criteria (including normal EEG background for age, at least 1 partial onset seizure, and unilateral or bilateral central/mid-temporal sharp waves with a positive horizontal dipole).

Age: The child's age is between 5 years, 0 months and 13 years, 11 months at study entry.

Language: The child must be a monolingual native speaker of English.

Handedness : The child must be right-handed.

Females: females of child bearing potential must agree to an acceptable and non-systemic form of birth control (including abstinence).

Intelligence: The child must have clinician-judged normal intelligence.

Academic History: The child must have an academic history of a regular education program (i.e., not in a special education class or program) without repeating grades.

Parent/Guardians:

* The patient's parent/guardian must be able to keep an accurate seizure record.
* Informed consent from the child's parent or legal guardian.
* Parents (guardians) must be able and willing to comply with instructions and study procedures.

Assent: Assent from the child if age 11 years or older.

Demographic characteristics: Children will be between 7 and < 14 years old at the time of enrollment. Children of both sexes and all race/ethnicities will be enrolled.

Exclusion Criteria for BECTS participants

Clinical Contraindications

* Children with diagnosis of Benign Occipital Epilepsy (BOE - normal EEG background, and unilateral or bilateral occipital sharp waves activated by eye closure).
* Children with history of primary generalized seizures (absence, myoclonic, drop).
* Children with mixed seizure disorder (e.g., Lennox-Gastaut Syndrome).
* Children sensory seizures only (i.e., auras).
* Children with diagnoses of pervasive developmental disorders (e.g., autism/autism spectrum disorders).
* Children with progressive neurological disease (e.g., degenerative, progressive neoplasm).
* Children with major medical disease (e.g., IDDM, depression, suicide attempt. cancer, renal failure).
* Children with a history of neonatal seizures.

Pregnancy: Children who are pregnant will not be eligible for enrollment.

Prior Therapy

* Children previously or currently treated with an AED for any reason (other than non chronic benzodiazepine, e.g., ED treatment).
* Children taking any psychoactive agent other than psychostimulants for ADD/ADHD.
* Children taking a psychostimulant for ADD/ADHD and not on a stable dose for at least 2 weeks at time of study enrollment.

MRI

• Standard MRI exclusion criteria, e.g. orthodontic braces, cochlear implant or other metallic implants which obscure or interfere with the MRI.

Special Education: Children with a special education placement based on ability or behavior.

Informed Consent: Inability or unwillingness of child or legal guardian/representative to give written informed consent.

Child not fluent in English.

Inclusion Criteria for Healthy Controls

Language: The child must be a monolingual native speaker of English.

Handedness: The child must be right-handed.

Females: Females of child bearing potential must agree to an acceptable and non-systemic form of birth control (including abstinence).

Intelligence: The child must have clinician-judged normal intelligence.

Academic History: The child must have an academic history of a regular education program (i.e., not in a special education class or program) without repeating grades.

Parents/Guardians:

* Informed consent from the child's parent or legal guardian.
* Parents (guardians) must be able and willing to comply with instructions and study procedures.

Assent: Assent from the child if age 11 years or older.

Demographic characteristics: Children will be between 5 and < 14 years old at the time of enrollment. Children of both sexes will be enrolled and no child will be excluded on the basis of race/ethnicity.

Exclusion Criteria for Healthy Controls

Clinical Contraindications

* Children with a diagnosis of a chronic neurological disorder.
* Children with diagnoses of pervasive developmental disorders (e.g., autism/autism spectrum disorders).
* Children with progressive neurological disease (e.g., degenerative, progressive neoplasm).
* Children with major medical disease (e.g., IDDM, cancer, renal failure).
* Children with a history of neonatal seizures.
* Pregnancy: Children who are pregnant will not be eligible for enrollment.

Prior Therapy

* Children previously or currently treated with an AED for any reason (other than non chronic benzodiazepine, e.g., ED treatment).
* Children taking any psychoactive agent other than psychostimulants for ADD/ADHD.
* Children taking a psychostimulant for ADD/ADHD and not on a stable dose for at least 2 weeks at time of study enrollment.

MRI and MRI/EEG Abnormality

• Standard MRI exclusion criteria, e.g. orthodontic braces, cochlear implant or other metallic implants which obscure or interfere with the MRI.

Special Education: Children with a special education placement based on ability or behavior.

Informed Consent: Inability or unwillingness of child or legal guardian/representative to give written informed consent.

Child not fluent in English.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of Centrotemporal Spikes per minute on EEG | 52 weeks

SECONDARY OUTCOMES:
Composite Score on CELF-4 Core Subtests (Language) | 52 Weeks
fMRI Lateralization indices for three language tasks | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Vannest, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Tenney JR, Glauser T, Altaye M, Szaflarski JP, Spencer C, Morita D, Vannest J. Longitudinal stability of interictal spikes in benign epilepsy with centrotemporal spikes. Epilepsia. 2016 May;57(5):805-11. doi: 10.1111/epi.13367. Epub 2016 Mar 25. PMID 27012680
- [Result] Vannest J, Tenney JR, Altaye M, Byars AW, Spencer C, Maloney TC, Szaflarski JP, Morita D, Glauser TA. Impact of frequency and lateralization of interictal discharges on neuropsychological and fine motor status in children with benign epilepsy with centrotemporal spikes. Epilepsia. 2016 Aug;57(8):e161-7. doi: 10.1111/epi.13445. Epub 2016 Jun 28. PMID 27350662